CLINICAL TRIAL: NCT01872429
Title: Short- and Long-Term Impact of Subtotal Parathyroidectomy on the Achievement of Bone and Mineral Parameters Recommended by Clinical Practice Guidelines in Dialysis Patients
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FEMH-IRB-102034-E
Record Dates: First submitted 2013-06-05; First posted 2013-06-07 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-04

CONDITIONS: Hyperparathyroidism
Keywords: subtotal parathyroidectomy; calcium; phosphorus; parathyroid hormone; hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Short-term group: Patients with postoperative 6-month laboratory data were included in the short-term group
- Long-term group: Patients with postoperative more than 6-month laboratory data were included in the long-term group

SUMMARY:
The impact of parathyroidectomy (PTX) on the bone mineral parameters in dialysis patients with secondary hyperparathyroidism (SHPT) remains unclear. The investigators performed this study to present the short- and long-term impact of PTX on calcium, phosphorus and intact parathyroid hormone control in dialysis patients with severe SHPT after operation. In particular, the investigators evaluate the impact based on the achievement of recommendations of the current clinical practice guidelines for bone and mineral parameters in dialysis patients after PTX.

DETAILED DESCRIPTION:
1. A retrospective chart review of dialysis patients including referred cases, receiving surgical PTX, which was performed by one surgeon at the Far Eastern Memorial Hospital, a 1084-bed tertiary-care medical center in northern Taiwan will be performed.
2. Serum levels of calcium, phosphorus and intact parathyroid hormone were routinely measured for three consecutive post-operative days and subsequent laboratory values were checked during out-patient follow-up period. Patients with postoperative 6-month laboratory data are included in the short-term group and those with more than 6-month available data are in the long-term one.
3. The National Kidney Foundation Kidney Disease Outcomes Quality Initiative (NKF-K/DOQI™) Clinical Practice Guidelines provided recommended target values for serum intact parathyroid hormone (iPTH)(150-300 pg/ml), phosphorus (3.5-5.5 mg/dl), calcium (8.4-9.5 mg/dl) and the calcium-phosphorus product (<55 mg2/dl2). The Kidney Disease: Improving Global Outcomes (KDIGO) Clinical Practice Guidelines suggested maintaining serum calcium in the reference range (8.5-10.5 mg/dl), phosphorus (2.7-4.5 mg/dl) and PTH values in the range of two to nine times the upper reference limit (130 - 585 pg/ml) in dialysis patients.
4. The investigators evaluated the impact of subtotal PTX on the control of bone and mineral parameters in dialysis patients with secondary HPT as the percentages of cases achieving the recommended K/DOQI and KDIGO targets.

ELIGIBILITY:
Inclusion Criteria:

* dialysis patients
* secondary hyperparathyroidism refractory to medical treatment
* patients receiving subtotal parathyroidectomy by one surgeon
* available laboratory data for at least six months after surgery

Exclusion Criteria:

* patients receiving parathyroidectomy other than subtotal type by other surgeon
* available laboratory data less than six months after surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dialysis patients, including referred cases, from the tertiary-care medical center in northern Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The percentages of cases achieving the recommended K/DOQI and KDIGO targets for bone mineral parameters after subtotal PTx | Twelve year period after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan